CLINICAL TRIAL: NCT06876961
Title: Effect of Arm Cycling Exercise on Pulmonary Functions After Colectomy In Elderly
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Israa Mohammed AbdelMoneim Youssef, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Israa-005640
Record Dates: First submitted 2025-03-07; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Function; Colectomy; Colorectal Cancer; Post-operative Rehabilitation; Intensive Care Unit (ICU) Acquired Weakness (ICU - AW); Arm Cycle Ergometer; Pulmonary Rehabilitation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm cycling exercise (Experimental): The study group, including 30 participants, will do 20 minutes of arm cycling exercise plus the traditional physical therapy program.
  Interventions: Other: Arm cycling exercise; Other: The traditional physical therapy program
- traditional physical therapy (Active Comparator): The control group, including 30 participants, will do the traditional physical therapy program only
  Interventions: Other: The traditional physical therapy program

INTERVENTIONS:
Other: Arm cycling exercise — The study involves a 20-minute arm cycling exercise twice daily for five days, starting with a warming-up and ending with a cooling-down. The workload is gradually increased to 60-70% of maximal heart rate, with patients sitting on a back support chair with 20 degrees backward inclination.
  Arms: Arm cycling exercise
Other: The traditional physical therapy program — The patient undergoes 10 minutes of deep diaphragmatic breathing exercises, 10 minutes of spirometer training, 3-set ankle pump and heel slide exercises, 10-minute sitting on the bed edge, 5 minutes of walking in the intensive care unit, and 3-set active free range of motion exercises.

SUMMARY:
This study will be done to investigate the effect of arm cycling on exercise and functional capacity, arterial blood gases, pulmonary functions, diaphragmatic excursion, time to peak inspiratory amplitude, physical function, anxiety, and depression after colectomy in the elderly.

DETAILED DESCRIPTION:
Around 42% of older patients with Chronic Respiratory Disease are considered 'frail', putting them at higher risk of adverse outcomes after surgery. Factors such as poor frailty, high comorbidity, low physical performance, poor nutritional state, or cognitive impairment increase the risk. Postoperative complications, such as pulmonary complications, can lead to increased morbidity, mortality, and hospital stays. Preoperative physiotherapy and exercise interventions have been suggested as preventive solutions. However, many patients undergo emergency surgery, emphasizing the need for strict postoperative care pathways. Exercise interventions, such as upper extremity aerobic exercise, have shown benefits in improving immobilization, oxygen consumption, ventilation, heart rate response, dyspnea, and quality of life. This study aims to investigate the effects of arm cycling on exercise capacity, arterial blood gases, pulmonary functions, diaphragmatic excursion, anxiety, and depression after colectomy in the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Sixty male patients who received a surgical removal of a diagnosed colon cancer (i.e., including right, transverse, left, sigmoid, subtotal, total, and hemicolectomy) will be included.
2. Patients with a histologically confirmed diagnosis of primary colon or rectal neoplasm.
3. Colectomy isolated surgeries.
4. Patients will be included in this study after the immediate admission to the intensive care unit.
5. The age of patients will be ≥ 65 years old.
6. Patients' body mass index will be < 30 Kg/m2.
7. All patients will be conscious, medically stable, and able to respond to the given commands fully.
8. Patients who voluntarily cooperated with this study
9. Karnofsky Performance Status > 60 and able to walk ≥ 60 m. The Karnosky Performance Status is one of the most used validated scales to define the functional status of a cancer patient. A Karnofsky Performance Status ≤ 60 indicates the inability to work and severe difficulty in carrying out activities of daily living and personal care of the cancer patient Before surgeries

Exclusion Criteria:

Men who will meet one of the following criteria will be excluded:

1. relapsing cancer or metastasis cancer; simultaneous diagnosis of other neoplasms.
2. Cardiac disease patients.
3. Chronic inflammatory autoimmune disease
4. Patients with neurological conditions limit the performance of exercises.
5. Patients with diagnosed psychogenic diseases.
6. Patients with musculoskeletal disorders that interfere with performing exercise programs.
7. Chronic obstructive pulmonary disease, Asthma, hemodynamically unstable, significant arrhythmias, and any chronic lung disease.
8. Patients require invasive/noninvasive ventilatory support.
9. regular use of immunosuppressive drugs.
10. Patients with cognitive disorders and unstable hemodynamics.
11. patients suffering from brain death; or respiratory failure; ventilator-dependent patients: patients receiving palliative care or patients on tracheostomy.
12. inability to understand given information due to language or intellectual barriers.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Sixty male patients who received a surgical removal of a diagnosed colon cancer (i.e., including right, transverse, left, sigmoid, subtotal, total, and hemicolectomy) will be included.
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Assessing the change of forced vital capacity using spirometry | At baseline and at the day 5 post-operative
  It will be conducted noninvasively using a spirometer, measuring: forced vital capacity (FVC) in Litres is known as total exhaled volume.
Assessment of change of functional capacity | At baseline and at the day 5 post-operative
  A 6-minute stepper test is proposed to evaluate exercise tolerance using a standardized protocol. The test measures the number of steps performed on a stepper in 6 minutes, equivalent to the 6-minute walk test. Patients are accustomed to the stepper for 2 minutes, followed by a 3-minute rest and 6-minute stepping period. Heart rate and oxygen saturation are monitored, and an investigator stays behind the patient throughout the test.
Assessment of change of diaphragmatic excursion using ultrasonography | At baseline and at the day 5 post-operative
  Participants undergo ultrasonography to measure diaphragmatic excursion In centimeters (cm) . The measurement will be performed using a 1- to 5-MHz ultrasound transducer in M-mode.
Assessment of change of diaphragmatic excursion using ultrasonography | At baseline and at the day 5 post-operative
  Participants undergo ultrasonography to measure the Time-to-peak inspiratory amplitude (TPIAdia) of the diaphragm during tidal breathing in seconds (sec) of each hemidaphragm ( right and left ). The measurement will be performed using a 1- to 5-MHz ultrasound transducer in M-mode.
Assessing the change of forced expiratory volume in 1 second using spirometry | At baseline and at the day 5 post-operative
  It will be conducted noninvasively using a spirometer, measuring:
  2-forced expiratory volume in 1 second (FVC1) in liters is known as volume exhaled in the first second.

SECONDARY OUTCOMES:
Assessment of change of potential of partial pressure of oxygen | At baseline and at the day 5 post-operative
  Arterial geometry will be used to examine the effect of cycling exercise on gas exchange, including the potential of partial pressure of oxygen (PaO₂) in millimeters of mercury (mmHg)
Assessment of change of bicarbonate (HCO₃) | At baseline and at the day 5 post-operative
  Arterial geometry will be used to examine the effect of cycling exercise on gas exchange, including the bicarbonate (HCO₃) in millimoles per liter (mmol/L)
Assessment of change of anxiety | At baseline and at the day 5 post-operative
  The Hospital Anxiety and Depression Scale will be used. it is a 14-item self-report screening scale with 7 items each for anxiety. A score of 0-7 is considered normal; 8-10 indicates mild illness, 11-15 moderate illness, and scores 16-21 are suggestive of severe illness
Assessment of change of depression | At baseline and at the day 5 post-operative
  The Hospital Anxiety and Depression Scale will be used. it is a 14-item self-report screening scale with 7 items each for depression. A score of 0-7 is considered normal; 8-10 indicates mild illness, 11-15 moderate illness, and scores 16-21 are suggestive of severe illness
Assessment of change of physical function in intensive care unit tested scored (PFIT) | At baseline and at the day 5 post-operative
  Physical function in intensive care test score (PFIT)-s will be used to assess physical function, consisting of four components: 1-assistance, 2-marching, 3-shoulder flexion strength, and 4-knee extension strength.
  The strength was based on the Oxford grading system, with each component mentioned above scoring 0-3 and summed to a maximum ordinal score of 12 points, Ranging from 0-12 with a higher score reflecting a better physical function.
Assessment of change of partial pressure of carbon dioxide (PaCO₂) | At baseline and at the day 5 post-operative
  Arterial geometry will be used to examine the effect of cycling exercise on gas exchange, including the partial pressure of carbon dioxide (PaCO₂) in millimeters of mercury (mmHg).
Assessment of change of potential of hydrogen (PH) | At baseline and at the day 5 post-operative
  Arterial geometry will be used to examine the effect of cycling exercise on gas exchange, including the potential of hydrogen (PH)
Assessment of change of lactate | At baseline and at the day 5 post-operative
  Arterial geometry will be used to examine the effect of cycling exercise on gas exchange, including the lactate millimoles per liter (mmol/L).

CONTACTS AND LOCATIONS:
Locations (1):
- the intensive care unit of King Hamad University Hospital,, Al Muharraq, Bahrain